CLINICAL TRIAL: NCT03313791
Title: Postprandial Blood Amino Acid Concentrations After Dairy Consumption
Brief Title: Postprandial Blood Amino Acid Response
Acronym: PARROT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL62458.072.17; NIZO175 (Other: NIZO)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Protein Digestion Kinetics
MeSH Terms: interventions — Whey; Yogurt; Mutation

STUDY DESIGN:
Intervention Model Description: 2 groups of 10 subjects both receive a different set of 6 different dairy products. Each subject within a group will receive all treatments on the same day of the week with a 1 week washout period between treatments. Results of the two groups will be analyzed separately, and products will only be compared within the same group of subjects, treating the data as two independent studies.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Whey protein concentrate (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Whey protein concentrate
- Yoghurt (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Yoghurt
- 50%whey-50% casein (Standard) (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: 50%whey-50% casein (Standard)
- 50%whey-50% casein (Alternative) (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: 50%whey-50% casein (Alternative)
- Micellar Casein Isolate- WPH (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Micellar Casein Isolate- WPH
- Micellar Casein Isolate - Na-caseinate (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Micellar Casein Isolate - Na-caseinate
- Micellar Casein Isolate (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Micellar Casein Isolate
- UHT milk (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: UHT milk
- Recombined milk (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Recombined milk
- Recombined 50% whey milk (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Recombined 50%whey milk
- Ca-caseinate (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Ca-caseinate
- Milk protein isolate (Experimental): portion size that contains 25 g of protein, oral, single administration
  Interventions: Dietary Supplement: Milk protein isolate

INTERVENTIONS:
Dietary Supplement: Whey protein concentrate — see arm description
  Arms: Whey protein concentrate
Dietary Supplement: Yoghurt — see arm description
  Arms: Yoghurt
Dietary Supplement: 50%whey-50% casein (Standard) — see arm description
  Arms: 50%whey-50% casein (Standard)
Dietary Supplement: 50%whey-50% casein (Alternative) — see arm description
  Arms: 50%whey-50% casein (Alternative)
Dietary Supplement: Micellar Casein Isolate- WPH — see arm description
  Arms: Micellar Casein Isolate- WPH
Dietary Supplement: Micellar Casein Isolate - Na-caseinate — see arm description
  Arms: Micellar Casein Isolate - Na-caseinate
Dietary Supplement: Micellar Casein Isolate — see arm description
  Arms: Micellar Casein Isolate
Dietary Supplement: UHT milk — see arm description
  Arms: UHT milk
Dietary Supplement: Recombined milk — see arm description
  Arms: Recombined milk
Dietary Supplement: Recombined 50%whey milk — see arm description
  Arms: Recombined 50% whey milk
Dietary Supplement: Ca-caseinate — see arm description
  Arms: Ca-caseinate
Dietary Supplement: Milk protein isolate — see arm description
  Arms: Milk protein isolate

SUMMARY:
This study was designed to obtain information about the change in postprandial amino acids in blood over time, after consumption of different dairy products with varying proportions of whey protein and caseins, and different processing conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65y
* BMI 18.5-30 kg/m2
* Non-smoking
* Healthy as assessed by the NIZO lifestyle and health questionnaire ("Verklaring leefgewoonten en gezondheid") and according to the judgment of the study physician.".
* Regular and normal Dutch eating habits as assessed by the NIZO lifestyle and health questionnaire (3 main meals per day)
* Veins suitable for cannulation (blood sampling)
* Voluntary participation
* Having given written informed consent
* Willing to comply with study procedures
* Accept use of all encoded data, including publication, and the confidential use and storage of all data for 15 years.
* Accept disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 30 days before Day 01 of this study
* Having a history of medical or surgical events that may significantly affect the study outcome, including: Inflammatory bowel disease, hepatitis, pancreatitis, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal disorders, colon or GI tract cancer
* Use of the following medication: glucose lowering drugs, insulin; medication that may impact gastric emptying (e.g. gastric acid inhibitors or laxatives)
* Diagnosed with diabetes, being treated for high blood glucose or increased fasting blood glucose (> 7 mmol/l in finger prick blood) as assessed during screening visit
* For men: Hb <8,5 mmol/l as assessed during screening visit; for women: Hb <7,5 mmol/l.
* Use of protein supplements
* Mental status that is incompatible with the proper conduct of the study
* A self-reported reported food allergy or sensitivity to dairy ingredients
* Alcohol consumption for men > 28 units/week and >4/day; for women: >21 units/week and >3/day
* Reported weight loss or weight gain of > 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period
* Reported slimming or medically prescribed diet
* Recent blood donation (<1 month prior to Day 01 of the study)
* Not willing or afraid to give up blood donation during the study
* Personnel of NIZO food research, FrieslandCampina Research, or Wageningen University, department of Human Nutrition, their partner and their first and second degree relatives
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results and eventual adverse events to and from his general practitioner
* Self reported pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
iAUC for postprandial individual plasma amino acids | Time Frame: 0-300 min after consumption
Cmax for postprandial individual plasma amino acids | Time Frame: 0-300 min after consumption

CONTACTS AND LOCATIONS:
Overall Officials: Alwine Kardinaal, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO, Ede, Netherlands